CLINICAL TRIAL: NCT06864182
Title: A Study to Evaluate the Relative Bioavailability of Single-Dose CX2101A Tablets and Enteric-Coated Tablets, and the Pharmacokinetics of Single and Multiple Doses of CX2101A Tablets in Healthy Adult Subjects
Brief Title: Relative Bioavailability Study of CX2101A for the Treatment of COVID-19
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Heronova Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SHRC-CX2101-01-02
Record Dates: First submitted 2025-02-24; First posted 2025-03-07 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: COVID-19; Coronavirus Infection
MeSH Terms: conditions — COVID-19; Coronavirus Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- CX2101A Placebo Tablet (Placebo Comparator): Participants from SAD cohort received single dose of CX2101A placebo tablet orally. Participant from MAD cohort received CX2101A placebo tablet orally once daily for 5 days.
  Interventions: Drug: CX2101A placebo enteric-coated tablet
- CX2101A Tablet (Experimental): Participants from SAD cohort received single dose of CX2101A tablet orally. Participant from MAD cohort received CX2101A tablet orally once daily for 5 days. Dose levels are 40 mg, 100mg, 160mg.
  Interventions: Drug: CX2101A tablet
- CX2101A Placebo Enteric-Coated Tablet (Placebo Comparator): Participants received single dose of CX2101A placebo enteric-coated tablet.
  Interventions: Drug: CX2101A placebo tablet
- CX2101A Enteric-Coated Tablet (Experimental): Participants received single dose of 100 mg CX2101A enteric-coated tablet.
  Interventions: Drug: CX2101A enteric-coated tablet

INTERVENTIONS:
Drug: CX2101A tablet — CX2101A tablet
  Arms: CX2101A Tablet
Drug: CX2101A placebo tablet — CX2101A placebo tablet
  Arms: CX2101A Placebo Enteric-Coated Tablet
Drug: CX2101A enteric-coated tablet — CX2101A enteric-coated tablet
  Arms: CX2101A Enteric-Coated Tablet
Drug: CX2101A placebo enteric-coated tablet — CX2101A placebo enteric-coated tablet
  Arms: CX2101A Placebo Tablet

SUMMARY:
The study comprises three parts: single ascending dose (SAD) studies of CX2101A tablets at 40 mg, 100 mg, and 160 mg; a relative bioavailability (BA) study comparing single-dose administration of 100 mg CX2101A tablets and enteric-coated tablets; and a multiple ascending dose (MAD) study of CX2101A tablets. The BA study (100 mg) is integrated into the SAD study(Nested within the SAD protocol to optimize resource utilization).

DETAILED DESCRIPTION:
1. Randomized, Double-Blind, Placebo-Controlled Design All studies are conducted under standardized fasting conditions to eliminate food interference Blinding is maintained throughout the entire study period for both subjects and investigators
2. Single Ascending Dose (SAD) Study Dose Groups: 40 mg, 100 mg, 160 mg (3 cohorts) Subject Allocation: 10 subjects/cohort (8 CX2101A + 2 placebo)

   Integration with BA Study:

   The 100 mg cohort will serve as the reference for bioavailability evaluation Subjects completing SAD phase will proceed to receive enteric-coated formulations
3. Multiple Ascending Dose (MAD) Study Dose Groups: Same 40 mg, 100 mg, 160 mg cohorts Subject Allocation: 10 subjects/cohort (8 CX2101A + 2 placebo) Administration Schedule: Daily dosing for 5 consecutive days Relative Bioavailability (BA) Study
4. Cohort Integration: Conducted within the 100 mg SAD group (N=10)

Treatment Sequence:

Initial single-dose administration of CX2101A tablets

≥7-day washout period (PK data-driven adjustment) Second single-dose administration of enteric-coated tablets

Subject Allocation:

CX2101A tablets group: 8 subjects (CX2101A + 8 placebo) Enteric-coated group: 8 subjects (CX2101A + 8 placebo)

ELIGIBILITY:
Inclusion Criteria:

1. Healthy volunteers aged between 18 and 55 years old (including 18 and 55 years old), regardless of gender.
2. For male volunteers, the body weight should be ≥ 50.0 kg, and for female volunteers, the body weight should be ≥ 45.0 kg. The body mass index (BMI) = body weight (kg) / height² (m²), and it should be within the range of 19.0 to 28.0 kg/m². Women of childbearing potential (WOCBP) or the female partners of male subjects should be willing to have no plans for childbearing from 2 weeks before the screening until 1 months after the last administration of the investigational medicinal product, and voluntarily adopt effective contraceptive measures (including one or more non-pharmacological contraceptive measures), and have no plans for sperm donation or egg donation.
3. No history of major diseases, and the results of physical examination, vital signs, 12-lead electrocardiogram, chest X-ray examination and laboratory tests during the screening period are normal, or although slightly beyond the normal reference value range, they are judged by the investigator to have no clinical significance.
4. The subject should be able to maintain good communication with the investigator, comply with various requirements of the clinical trial, and voluntarily sign the informed consent form.

Exclusion Criteria:

1. Diseases with abnormal clinical manifestations that occurred before screening or are currently occurring and need to be excluded, including but not limited to those in the nervous/mental system, respiratory system, cardiovascular and cerebrovascular system, digestive system (any history of gastrointestinal diseases that affect drug absorption), hematological and lymphatic system, urinary system, endocrine system, and immune system.
2. Acute diseases that occurred from the screening stage to before the first administration of the investigational medicinal product and are judged by the investigator to possibly affect the research results.
3. Subjects who cannot tolerate intravenous puncture or those with a history of syncope judged by the investigator to be of clinical significance.
4. Subjects with difficulty in swallowing.
5. Subjects who are judged by the investigator to possibly or definitely have an allergic reaction to the investigational drug (including similar drugs), or any of its excipients; or subjects with an allergic constitution judged by the investigator to be of clinical significance (a history of severe allergies to multiple drugs and foods) or a history of allergic diseases.
6. Subjects who have undergone surgery before screening and are judged by the investigator to possibly affect the absorption, distribution, metabolism, and excretion of the drug, or subjects with severe surgical sequelae, or subjects who plan to undergo surgery during the study period.
7. Subjects who donated blood or had massive blood loss (≥ 400 mL), donated ≥ 2 units of component blood, or received a blood transfusion within 3 months before screening, or those who plan to donate blood during the trial.
8. Subjects who received any investigational drug in a clinical study or participated in any interventional clinical study within 3 months before screening.
9. Subjects who smoked an average of more than 5 cigarettes per day within 3 months before screening, or those who cannot stop using any tobacco products during the trial.
10. Subjects who consumed an average of more than 14 units of alcohol per week within 3 months before screening (1 unit of alcohol ≈ 360 mL of beer or 45 mL of spirits with an alcohol content of 40% or 150 mL of wine), or those who cannot stop using any alcohol-containing products during the trial, or those with a positive alcohol breath test before the administration of the trial.
11. Subjects who consumed an excessive amount of tea, coffee, and/or caffeine-containing beverages on average per day (more than 8 cups on average, 1 cup ≈ 250 mL) within 3 months before screening, or those who cannot stop consuming tea, coffee, and/or caffeine-containing beverages during the trial.
12. Subjects who used any prescription drugs, over-the-counter drugs, traditional Chinese patent medicines, Chinese herbal medicines, vitamins, or health foods within 28 days before screening or within 5 drug half-lives (whichever is longer).
13. Female subjects who are pregnant or breastfeeding, or those with a positive blood/urine pregnancy test (only for WOCBP) at any time during screening.
14. Positive results or results exceeding the upper limit of the reference range for the four hemodialysis tests: hepatitis B surface antigen (HBsAg), quantitative hepatitis C (HCV) antibody, quantitative human immunodeficiency virus (HIV) antibody, or treponema pallidum antibody.
15. Subjects with a positive urine drug screening (morphine, tetrahydrocannabinolic acid, methamphetamine, methylenedioxymethamphetamine, ketamine) or those with a history of drug abuse or drug use within the past 5 years before the trial.
16. Subjects who consumed or drank pitaya, mango, pomelo, carambola, or foods or beverages prepared from them, or foods or beverages containing xanthine, caffeine, or alcohol (including chocolate, tea, coffee, cola, cocoa, etc.), or other special diets that affect the absorption, distribution, metabolism, and excretion of the drug within 72 hours before screening.
17. Subjects with special dietary requirements, lactose intolerance, those without a habit of eating breakfast, or those who cannot accept the unified diet.
18. Subjects who, according to the investigator's judgment, are not suitable to participate in this trial.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2024-03-21 (Actual); Primary Completion 2024-05-25 (Actual); Study Completion 2024-05-25 (Actual)

PRIMARY OUTCOMES:
PK profile of CX2101A and its metabolite CX210101 and CX210108 | From time zero up to 96 hours post-dose following last dose of CX2101A
  Peak Concentration (Cmax): The maximum plasma concentration of the drug.
PK profile of CX2101A and its metabolite CX210101 and CX210108 | From time zero up to 96 hours post-dose following last dose of CX2101A
  Area Under the Curve from Time Zero to the Last Measurable Concentration (AUC0-t): The area under the plasma concentration-time curve from time zero to the last measurable concentration.
PK profile of CX2101A and its metabolite CX210101 and CX210108 | From time zero up to 96 hours post-dose following last dose of CX2101A
  Area Under the Curve from Time Zero Extrapolated to Infinity (AUC0-∞): The area under the plasma concentration-time curve from time zero extrapolated to infinity.
PK profile of CX2101A and its metabolite CX210101 and CX210108 | From time zero up to 96 hours post-dose following last dose of CX2101A
  Time to Reach Peak Concentration (Tmax): The time at which the peak plasma concentration is reached.
PK profile of CX2101A and its metabolite CX210101 and CX210108 | From time zero up to 96 hours post-dose following last dose of CX2101A
  Elimination Half-Life (T1/2): The time required for the plasma concentration to decrease by half.
PK profile of CX2101A and its metabolite CX210101 and CX210108 | From time zero up to 96 hours post-dose following last dose of CX2101A
  Apparent Volume of Distribution (Vz/F): The volume into which the drug appears to be distributed, corrected for bioavailability.
PK profile of CX2101A and its metabolite CX210101 and CX210108 | From time zero up to 96 hours post-dose following last dose of CX2101A
  Apparent Clearance (CL/F): The clearance of the drug from the plasma, corrected for bioavailability.
PK profile of CX2101A and its metabolite CX210101 and CX210108 | From time zero up to 96 hours post-dose following last dose of CX2101A
  Percentage of AUC Extrapolated (AUC_%Extrap): The percentage of the total AUC that is extrapolated beyond the last measurable concentration.

SECONDARY OUTCOMES:
Rate and severity of treatment-emergent adverse events (TEAEs) | From day 1 until 4 days after treatment
  Based on the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version 5.0
Vital signs | From day 1 until 4 days after treatment
  Number of participants with abnormal results of vital signs.
Electrocardiogram (ECG) | From day 1 until 4 days after treatment
  Number of participants with abnormal results of electrocardiogram.
Physical examinations | From day 1 until 4 days after treatment
  Number of participants with abnormal results of physical examinations
Complete blood count test | From day 1 until 4 days after treatment
  Number of participants with abnormal results of complete blood count test.
Clinical Chemistry | From day 1 until 4 days after treatment
  Number of participants with abnormal results of clinical chemistry.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang Xiaoshan Hospital, Hangzhou, China

IPD SHARING:
Plan to Share IPD: No